CLINICAL TRIAL: NCT06696703
Title: Effect of Human Urinary Kallidinogenase on Inflammatory Factors in Acute Ischemic Stroke: a Single-center, Randomized, Open Label, Blinded-endpoint, Controlled Study(KIF-AIS)
Brief Title: Effect of Human Urinary Kallidinogenase on Inflammatory Factors in Acute Ischemic Stroke (KIF-AIS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Zhongling Zhang, Doctor, First Affiliated Hospital of Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023155
Record Dates: First submitted 2024-11-16; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; Urinary Kallidinogen; Inflammatory factors; 90 days functional outcomes
MeSH Terms: conditions — Ischemic Stroke | interventions — Injections; Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human Urinary Kallidinogenase for injection (HUK) (Experimental): Patients in this arm will be given urinary kallidinogenase for injection，0.15 peptide nucleic acids (PNA)， once a day for 7days plus routine clinical treatment
  Interventions: Drug: Human urinary kininogenase(HUK)
- sham-HUK treatment (Placebo Comparator): Normal sodium chloride injection plus routine clinical treatment
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Human urinary kininogenase(HUK) — Experimental group (HUK plus routine clinical treatment): administered within 48 hours of AIS onset, 0.15PNA unit was dissolved in 100ml sodium chloride injection by intravenous infusion for not less than 50 minutes, once a day.
  Other Names: Urinary Kallidinogenase for Injection,Guangdong Tianpu Biochemical Pharmaceutical Co., Ltd, National Pharmaceutical Approval Letter H20052065
  Arms: Human Urinary Kallidinogenase for injection (HUK)
Other: Placebo — Placebo group (Normal sodium chloride injection plus routine clinical treatment): Normal sodium chloride administered within 48 hours of AIS onset, by intravenous infusion for not less than 50 minutes, once a day.
  Other Names: Normal sodium chloride injection
  Arms: sham-HUK treatment

SUMMARY:
The goal of this clinical trial is to explore the changes in the expression levels of inflammatory factors before and after the early treatment of Human Urinary Kallidinogen (HUK) in the acute ischemic stroke. It will also learn about the correlation between inflammatory factors and AIS prognosis, in order to clarify the efficacy and safety of Urinary Kallidinogen in the acute phase of AIS.

DETAILED DESCRIPTION:
The study process lasts for a total of 90 days, including the screening period, treatment period, and follow-up period. During the treatment period, the experimental group is treated with HUK in the 48 hours of AIS plus routine clinical treatment, while the control group receives routine clinical treatment group for 7 days.All patients are followed up until the 90th day after stroke. The sample size of the study is 200 patients. The ratio of the experimental group to the control group was 1:1.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis as acute ischemic stroke according to the Chinese guidelines for diagnosis and treatment of acute ischemic stroke 2018;
2. First clinical onset or previous presence of cerebral infarction without severe sequelae（Premorbid mRS ≤2）
3. Age≥18 years, male or female;
4. 3≤Baseline NIHSS≤25;
5. Written informed consent obtained from the patient or legally responsible person.

Exclusion Criteria:

1. Cerebral hemorrhage and the acute phase of other hemorrhagic diseases；
2. Previously allergic or intolerant to injectable HUK；
3. Used ACEI drugs prior to medication and less than 5 half-lives of the drug (according to the specific drug instructions) or received ACEI drugs during the study period;
4. Stent surgery after the AIS onset or planned interventional therapy;
5. Pregnancy, lactation or planned pregnancy；
6. Life expectancy of less than 3months or inability to complete the study for other reasons；
7. Unwilling to be followed up or poor compliance；
8. Current participation in other clinical research;
9. Other causes of AIS (such as dissection, vasculitis, pre-thrombotic lesions, drug abuse).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The Favorable Stroke Outcome of 90 days | 90 days after treatment
  mRS 0-2
The changes of the serum inflammatory markers before and after treatment | Baseline、1 day after treatment、3 days after treatment、90 days after treatment
  Complete Blood Count、CRP、IL-6、HCY、NSE

SECONDARY OUTCOMES:
The changes of NIHSS before and after treatment | Baseline、7 days after treatment
  National Institute of Health stroke scale, NIHSS
Stroke recurrence rate | 90 days after treatment
  Ischemic stroke
The incidence of intracranial hemorrhage | 90 days after treatment
  Symptomatic intracranial hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Zhongling Zhang, Principal Investigator — First Affiliated Hospital, Harbin Medical University
Locations (1):
- Zhongling Zhang, Harbin, Heilongjiang, China